CLINICAL TRIAL: NCT00379964
Title: A Noncomparative, Multicenter, Open-Label, Study to Evaluate the Safety, Tolerability and Efficacy of MK0991 as Empirical Therapy in Indian Adults With Persistent Fever and Neutropenia
Brief Title: A 28 - 90 Days Study to Evaluate the Safety, Tolerability, and Efficacy of Caspofungin Injection as Empirical Therapy in Indian Adults With Persistent Fever and Neutropenia (0991-053)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-053; 2006_037
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

INTERVENTIONS:
Drug: caspofungin acetate — Cancidas 50 mg dose followed by 70 mg load on day 1 was administered in Indian adults with persistent fever and neutropenia for a maximum duration of empirical treatment from 28 days ((for patients without documented infection) to 90 days (for patients with documented baseline or emergent fungal infection). Patients were treated until the resolution of neutropenia (ANC>500/mm3), and for up to 72 hours later.
  Other Names: MK0991; Cancidas

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of ertapenem sodium as initial therapy for the treatment of complicated urinary tract infections, including pyelonephritis in indian adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a low white cell count (less than 500/mm3) for at least 96 hours
* Patient is indian and is greater than 18 years of age
* Patient received chemotherapy for blood disorders and blood cancers

Exclusion Criteria:

* Patient has an invasive fungal infection
* Patient has a bacterial infection that is not controlled
* Patient has allergy to the class of antifungals of study drug
* Patient is not expected to survive at least 5 days
* Patient is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Any clinical or laboratory serious drug-related adverse experience during the study drug therapy period plus 14 days posttherapy. | during the study drug therapy period plus 14 days posttherapy

SECONDARY OUTCOMES:
Survival for at least 7 days following study therapy reduce fever during period of low white blood cell counts fungal infection no longer present following study therapy | 7 days following study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html